CLINICAL TRIAL: NCT02281552
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Phase 3 Study To Demonstrate Non-inferiority For The Efficacy Of A Once Daily Dose Of Tofacitinib Modified Release Tablet To A Twice Daily Dose Of The Immediate Release Tablet In Adult Patients With Rheumatoid Arthritis On Background Methotrexate
Brief Title: A Study To Evaluate The Safety And Efficacy Of Tofacitinib Modified Release Tablets Compared To Tofacitinib Immediate Release Tablets In Adult Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921215; TOFACITINIB QD P3 (Other: Alias Study Number)
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Tofacitinib, CP-690,550, Janis kinase, JAK inhibitor, modified release, Xeljanz
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tofacitinib modified release tablet (Experimental)
  Interventions: Drug: Tofacitinib
- tofacitinib immediate release tablet (Active Comparator)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — tofacitinib modified release 11 mg tablet administered once time a day for 12 weeks
  Arms: tofacitinib modified release tablet
Drug: Tofacitinib — tofacitinib immediate release 5 mg tablet administered twice a day for 12 weeks
  Arms: tofacitinib immediate release tablet

SUMMARY:
This is a 12 week study that will evaluate the efficacy and safety of the 11 mg tofacitinib modified release tablet taken once a day in patients with rheumatoid arthritis who continue taking methotrexate. Results for the modified release tablets will be compared to the efficacy and safety of the 5 mg tofacitinib immediate release tablets taken twice a day in patients with rheumatoid arthritis who continue taking methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rheumatoid arthritis
* currently taking a stable dose of methotrexate
* no evidence of active or latent or inadequately treated tuberculosis

Exclusion Criteria:

* evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic disease
* clinically significant infections within the past 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- Japan (36):
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - Yamada Rheumatology Clinic, Matsuyama, Ehime
  - St. Mary's Hospital, Kurume, Fukuoka
  - Gunma Rheumatism Clinic, Takasaki-shi, Gunma
  - Inoue Hospital, Tohrimachi, Takasaki, Gunma
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Katayama Orthopaedic Rheumatology Clinic, Asahikawa, Hokkaido
  - Yoshida orthopaedics and rheumatologyclinic, Morioka, Iwate
  - Komagamine Rheumatoid Orthopaedic Clinic, Morioka, Iwate
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Osaki Citizen Hospital, Oosaki, Miyagi
  - Tohoku University Hospital/ Department of Hematology and Rheumatology, Sendai, Miyagi
  - Nagano Red Cross Hospital, Nagano, Nagano
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - National Hospital Organization Ureshino Medical Center, Ureshino-shi, Saga-ken
  - Soshigayaokura clinic, Setagaya-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Honjo Rheumatism Clinic, Takaoka-shi, Toyama
  - Miyasato Clinic, Shūnan, Yamaguchi
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Sugimoto rheumatology and internal medicine clinic, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - SHONO Rheumatism Clinic, Fukuoka
  - Sagawa Akira Rheumatology Clinic, Hokkaido
  - Matsubara Mayflower Hospital, Hyōgo
  - Yokohama Minami Kyosai Hospital, Kanagawa
  - Kumamoto Orthopaedic Hospital, Kumamoto
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto
  - Oribe Clinic of Rheumatology and Internal Medicine, Ōita
  - Otsuka Clinic of Rheumatism and Medicine, Ōita
  - Rabbit Clinic, Saitama
  - Hirose Clinic, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Tanaka Y, Sugiyama N, Toyoizumi S, Lukic T, Lamba M, Zhang R, Chen C, Stock T, Valdez H, Mojcik C, Fan H, Deng C, Yuasa H. Modified- versus immediate-release tofacitinib in Japanese rheumatoid arthritis patients: a randomized, phase III, non-inferiority study. Rheumatology (Oxford). 2019 Jan 1;58(1):70-79. doi: 10.1093/rheumatology/key250. PMID 30137547
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921215&StudyName=A%20study%20to%20evaluate%20the%20safety%20and%20efficacy%20of%20tofacitinib%20modified%20release%20tablets%20compared%20to%20tofacitinib%20immediate%20release%20tablets%20in

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib Modified Release (MR): Participants orally received 11 milligrams (mg) of tofacitinib MR tablets once daily and matching placebo of tofacitinib IR tablets twice daily for 12 weeks.
- Tofacitinib Immediate Release (IR): Participants orally received 5 mg of tofacitinib IR tablets twice daily and matching placebo of tofacitinib MR tablets once daily for 12 weeks.
Period: Overall Study
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Started | 104 | 105
Completed | 100 | 95
Not Completed | 4 | 10
Not completed — Medication error | 1 | 0
Not completed — Insufficient clinical response | 0 | 1
Not completed — Adverse Event | 3 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized and received at least one dose of the randomized investigational drug.
Groups:
- Tofacitinib Modified Release (MR): Participants orally received 11 mg of tofacitinib MR tablets once daily and matching placebo of tofacitinib IR tablets twice daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR) | Total
Number analyzed (Participants) | 104 | 105 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.4) | 58.9 (10.2) | 58 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 75 | 161
  Male | 18 | 30 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 104 | 105 | 209
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score in 28 Joints Using 4 Variables (DAS28-4) (C-Reactive Protein [CRP]) at Week 12
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joints count, CRP (milligrams per liter [mg/L]) and patient global assessment of disease activity on a 100 millimeter (mm) visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (CRP) [less than or equal to] <= 3.2 implied low disease activity and greater than (>) 3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (CRP) less than (<) 2.6 implied remission.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all participants who were randomized and received at least one dose of the randomized investigational drug. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 100 | 95
units on a scale | -2.43 (0.09) | -2.85 (0.09)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) vs Tofacitinib Immediate Release (IR); Analysis was conducted using a linear mixed effect model with repeated measures (MMRM), which included treatment (tofacitinib MR 11 mg QD and IR 5 mg BID), visit, and treatment by visit interaction as fixed effects and participants as a random effect; Test type: Non-Inferiority — Non-inferiority of tofacitinib MR 11 mg QD to IR 5 mg BID was concluded if the upper bound of the 2-sided 95% confidence interval of differences between the treatment groups (MR 11 mg QD - IR 5 mg BID) at Week 12 was less than the pre-specified non-inferiority margin of 0.6; Least Square (LS) mean difference = 0.43, 95% CI 2-sided [0.17 to 0.69], Standard Error of Mean 0.13

2. Secondary Outcome: Change From Baseline in Disease Activity Score in 28 Joints Using 4 Variables (DAS28-4) (Erythrocyte Sedimentation Rate [ESR]) at Week 12
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (millimeters per hour [mm/hr]) and patient global assessment of disease activity on a 100 mm visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) <2.6 implied remission.
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized and received at least one dose of the randomized investigational drug. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this specified outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 99 | 95
units on a scale | -2.50 (0.09) | -2.86 (0.09)

3. Secondary Outcome: Number of Participants Achieving an American College of Rheumatology 20 Percent [%] (ACR20) Response at Week 12
Description: Participants with 20% improvement in 68-tender and 66-swollen joint counts and 20% improvement in at least 3 of the 5 measures: patient's global assessment of arthritis, physician global assessment of arthritis, patient's assessment of arthritis pain, health assessment questionnaire-disability index(HAQ-DI) and CRP. Patient's global assessment of arthritis: participant assessed arthritis by 100 mm VAS, score: 0 mm (no arthritis) to 100 mm (extreme arthritis), higher score implied more arthritis. Physician global assessment of arthritis: physician judged participants arthritis by 100 mm VAS, score: 0 mm (no arthritis) to 100 mm (extreme arthritis), higher score implied more arthritis. Patient's assessment of arthritis pain: participant assessed arthritis pain by 100 mm VAS, score: 0 mm (no pain) to 100 mm (most severe pain), higher score implied more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability.
Time Frame: Week 12
Population: FAS included all participants who were randomized and received at least one dose of the randomized investigational drug. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this specified outcome measure. Missing values due to withdrawal were imputed using non-responder imputation (NRI) method.
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 87 | 83

4. Secondary Outcome: Number of Participants Achieving an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants with 50% improvement in 68-tender and 66-swollen joint counts and 50% improvement in at least 3 of the 5 measures: patient's global assessment of arthritis, physician global assessment of arthritis, patient's assessment of arthritis pain, health assessment questionnaire-disability index(HAQ-DI) and CRP. Patient's global assessment of arthritis: participant assessed arthritis by 100 mm VAS, score: 0 mm (no arthritis) to 100 mm (extreme arthritis), higher score implied more arthritis. Physician global assessment of arthritis: physician judged participants arthritis by 100 mm VAS, score: 0 mm (no arthritis) to 100 mm (extreme arthritis), higher score implied more arthritis. Patient's assessment of arthritis pain: participant assessed arthritis pain by 100 mm VAS, score: 0 mm (no pain) to 100 mm (most severe pain), higher score implied more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability.
Time Frame: Week 12
Population: FAS included all participants who were randomized and received at least one dose of the randomized investigational drug. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this specified outcome measure. Missing values due to withdrawal were imputed using NRI method.
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 70 | 71

5. Secondary Outcome: Number of Participants Achieving an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants with 70% improvement in 68-tender and 66-swollen joint counts and 70% improvement in at least 3 of the 5 measures: patient's global assessment of arthritis, physician global assessment of arthritis, patient's assessment of arthritis pain, health assessment questionnaire-disability index(HAQ-DI) and CRP. Patient's global assessment of arthritis: participant assessed arthritis by 100 mm VAS, score: 0 mm (no arthritis) to 100 mm (extreme arthritis), higher score implied more arthritis. Physician global assessment of arthritis: physician judged participants arthritis by 100 mm VAS, score: 0 mm (no arthritis) to 100 mm (extreme arthritis), higher score implied more arthritis. Patient's assessment of arthritis pain: participant assessed arthritis pain by 100 mm VAS, score: 0 mm (no pain) to 100 mm (most severe pain), higher score implied more pain. HAQ-DI: functional disability evaluation, score: 0 (no difficulty) to 3 (extreme difficulty), higher score implied more disability.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 32 | 48

6. Secondary Outcome: Number of Participants With DAS Remission (DAS28-4-CRP <2.6) at Week 12
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from SJC and TJC using 28 joints count, CRP (mg/L) and patient global assessment of disease activity on a 100 mm visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (CRP) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (CRP) <2.6 implied remission. Number of participants with DAS remission (DAS28-4-CRP<2.6) were reported in this outcome measure.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 52 | 72

7. Secondary Outcome: Number of Participants With DAS Remission (DAS28-4-ESR <2.6) at Week 12
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hr) and patient global assessment of disease activity on a 100 mm visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) <2.6 implied remission. Number of participants with DAS remission (DAS28-4-ESR<2.6) were reported in this outcome measure.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 18 | 36

8. Secondary Outcome: Number of Participants With Low Disease Activity (DAS28-4-CRP <=3.2) at Week 12
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (CRP) was calculated from SJC and TJC using 28 joints count, CRP (mg/L) and patient global assessment of disease activity on a 100 mm visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (CRP) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (CRP) <2.6 implied remission. Number of participants with low disease activity (DAS28-4-CRP<=3.2) were reported in this outcome measure.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 76 | 82

9. Secondary Outcome: Number of Participants With Low Disease Activity (DAS28-4-ESR <=3.2) at Week 12
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28-4 (ESR) was calculated from SJC and TJC using 28 joints count, ESR (mm/hr) and patient global assessment of disease activity on a 100 mm visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition). Total DAS28-4 (ESR) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity. DAS28-4 (ESR) <=3.2 implied low disease activity and >3.2 to <=5.1 implied moderate disease activity, >5.1 implied high disease activity, and DAS28-4 (ESR) <2.6 implied remission. Number of participants with low disease activity (DAS28-4-ESR<=3.2) were reported in this outcome measure.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 44 | 63

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 categories of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities over past week. Each activity category consisted of 2-3 items. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 99 | 95
units on a scale | -0.44 (0.04) | -0.46 (0.04)

11. Secondary Outcome: Number of Participants Achieving an Improvement of at Least 0.22 Units in Health Assessment Questionnaire (HAQ Scores) at Week 12
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 categories of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities over past week. Each activity category consisted of 2-3 items. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities. Number of participants with an improvement of at least 0.22 units in HAQ scores from baseline to Week 12 were reported in this outcome measure.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 103 | 104
participants | 65 | 60

12. Secondary Outcome: Change From Baseline in the Short Form 36 (SF-36) Health Survey Domain Scores at Week 12
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: physical functioning, role physical, bodily pain, social functioning, mental health, role emotional, vitality, and general health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of 8 health aspects were aggregated to derive the two component scores (physical component scores [PCS], mental component scores [MCS]) ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 99 | 95
units on a scale
  Physical Functioning | 5.54 (0.67) | 6.29 (0.68)
  Role Physical | 6.51 (0.81) | 6.97 (0.83)
  Bodily Pain | 9.41 (0.77) | 11.92 (0.78)
  General Health | 4.53 (0.52) | 4.72 (0.53)
  Vitality | 8.07 (0.75) | 8.20 (0.76)
  Social Function | 4.26 (0.63) | 5.06 (0.64)
  Role Emotional | 7.23 (0.86) | 6.56 (0.87)
  Mental Health | 4.46 (0.80) | 5.26 (0.81)

13. Secondary Outcome: Change From Baseline in the Short Form 36 (SF-36) Health Survey Component Scores at Week 12
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: physical functioning, role physical, bodily pain, social functioning, mental health, role emotional, vitality, and general health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of 8 health aspects were aggregated to derive the two component scores PCS and MCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 99 | 95
units on a scale
  PCS | 6.59 (0.58) | 7.85 (0.59)
  MCS | 5.29 (0.76) | 5.08 (0.77)

14. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Scores at Week 12
Description: The FACIT-Fatigue Scale was a participant completed questionnaire consisted of 13 items that assessed fatigue. Each item was scored on a scale of 0 (not at all) to 4 (very much), Total score ranging from 0 (not at all) to 52 (very much), higher scores represented lower level of fatigue.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 99 | 95
units on a scale | 5.28 (0.66) | 6.12 (0.67)

15. Secondary Outcome: Change From Baseline in the European Quality of Life - 5 Dimensions Questionnaire (EQ-5D) Scores at Week 12
Description: EQ-5D was a participant completed instrument designed to assess impact on quality of life in terms of a single utility score in five domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression with 3 possible answers for each item (1=no problem, 2=moderate problems, 3=severe problems). The 5-dimensional systems are converted into a single index utility score between 0 and 1, where higher score indicated a better health state.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 99 | 95
units on a scale | 0.20 (0.02) | 0.25 (0.02)

16. Other Pre Specified Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events between first dose of study drug and up to 12 weeks that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non- serious adverse events.
Time Frame: Baseline up to 12 weeks
Population: Safety analysis set included all participants who were randomized and received at least one dose of the randomized investigational drug.
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 104 | 105
participants
  AEs | 55 | 54
  SAEs | 5 | 4

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Criteria: lipids(cholesterol[CH] milligrams/deciliter[mg/dL] >1.3*upper limit normal(ULN), high-density lipoprotein CH mg/dL <0.8*lower limit normal(LLN), Low-density lipoprotein CH mg/dL >1.2* ULN, triglycerides mg/dL >1.3*ULN); neutrophil count(NC) <1000 cells/cubic milliliters(mm^3), platelet counts(PC) <100,000 P/mm^3, lymphocyte counts(LC) <500 L/mm^3, any single (aspartate transaminase elevation(ASTE)/alanine transaminase elevation(ALTE) >=3*ULN, hemoglobin(Hb) value <8.0 grams(g)/dL or >=2 g/dL below baseline, any serum creatinine(SC) increase(inc) >50% or inc >0.5 mg/dL over the average of screening(OAS) and baseline values(BV), 2 sequential ASTE/ALTE>=3*ULN with total bilirubin value(TBV) >=2*ULN, ASTE/ALTE >=3*ULN, ASTE/ALTE >=5*ULN, Hb <8.0 g/dL or decrease of >30% from BV, PC <75,000 P/mm^3, NC <1000 cells/mm^3, LC <500 L/mm^3, confirmed inc in SC >50% OAS and BV and detection of hepatitis B virus-deoxyribonucleic acid(HBV-DNA) by the two sequential quantitative tests.
Time Frame: Baseline up to 12 weeks
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
Number analyzed (Participants) | 104 | 105
participants
  Cholesterol | 11 | 8
  High-density lipoprotein Cholesterol | 1 | 1
  Low-density lipoprotein Cholesterol | 22 | 21
  Triglycerides | 6 | 10
  Neutrophil counts <1000 cells/mm3 | 0 | 0
  Platelet counts <100,000 platelets/mm3 | 0 | 0
  Lymphocyte counts <500 lymphocytes/mm3 | 1 | 0
  Any single AST and/or ALT elevation >=3xULN | 1 | 0
  Any single Hb value <8.0 g/dL or >=2 gm/dL | 0 | 2
  Any serum creatinine increase >50% | 0 | 0
  2sequential AST/ALT elevations>=3xULN, TBV>=2xULN | 0 | 0
  2 sequential AST or ALT elevations >=3xULN | 1 | 0
  2 sequential AST or ALT elevations >=5xULN | 0 | 0
  2sequential Hb<8.0 g/dL or decrease of >30%from BV | 0 | 1
  2 sequential platelet counts <75,000 platelets/mm3 | 0 | 0
  2 sequential neutrophil counts <1000 cells/mm3 | 0 | 0
  2 sequential lymphocyte count <500 lymphocytes/mm3 | 0 | 0
  Confirmed increases in serum creatinine >50% | 0 | 0
  Detection of HBV-DNA | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 12 weeks
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety data set included all participants who received at least one dose of the study drug.
Arm/Group | Tofacitinib Modified Release (MR) | Tofacitinib Immediate Release (IR)
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/105
Serious Adverse Events (participants affected / at risk) | 5/104 | 4/105
Other Adverse Events (participants affected / at risk) | 10/104 | 13/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Modified Release (MR) (N=104) | Tofacitinib Immediate Release (IR) (N=105)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib Modified Release (MR) (N=104) | Tofacitinib Immediate Release (IR) (N=105)
Nasopharyngitis (Infections and infestations) | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02281552/SAP_000.pdf
  • Study Protocol (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02281552/Prot_001.pdf